CLINICAL TRIAL: NCT00008281
Title: A Multicenter, Open-Label, Randomized, Three-Arm Study Of 5-Fluorouracil (5-FU) Plus Leucovorin (LV) Or Oxaliplatin Or A Combination Of (5-Fu) LV + Oxaliplatin As Second-Line Treatment Of Metastatic Colorectal Carcinoma
Brief Title: Comparison of Three Chemotherapy Regimens in Treating Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sanofi (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068394; SANOFI-EFC4584; BRCC-00036
Record Dates: First submitted 2001-01-06; First posted 2004-02-16 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2002-04

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which regimen of chemotherapy is more effective for metastatic colorectal cancer.

PURPOSE: Phase III trial to compare the effectiveness of three chemotherapy regimens in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival of patients with metastatic colorectal carcinoma treated with fluorouracil and leucovorin calcium with vs without oxaliplatin vs oxaliplatin alone. II. Compare the response rate, time to tumor-related symptomatic worsening, time to disease progression, onset and duration of complete and partial responses, and duration of disease stabilization in patients treated with these regimens. III. Determine the safety profile of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to Karnofsky performance status (50-60% vs 70-100%), number of metastatic organs (1 vs 2 or more), and LDH value (up to 1.5 times upper limit of normal (ULN) vs greater than 1.5 times ULN). Patients are randomized to one of three treatment arms. Arm I: Patients receive leucovorin calcium IV over 2 hours followed by fluorouracil IV continuously over 22 hours on days 1 and 2. Arm II: Patients receive oxaliplatin IV over 2 hours on day 1. Arm III: Patients receive oxaliplatin IV concurrently with leucovorin calcium IV over 2 hours followed by fluorouracil IV continuously over 22 hours on day 1. Leucovorin calcium and fluorouracil are administered alone on day 2 on the same schedule as on day 1. Treatment repeats every 2 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients are followed for 30 days, every 2 weeks for up to 3 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 786 patients (262 per arm) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic adenocarcinoma of the colon or rectum that is not amenable to potentially curative therapy (e.g., inoperable metastatic disease) At least 1 unidimensionally measurable lesion at least 20 mm in diameter by conventional CT or MRI scan or at least 10 mm in diameter by spiral CT scan Progressive disease by CT or MRI scan during or no more than 6 months after the last dose of prior first-line irinotecan, fluorouracil, and leucovorin calcium (Saltz regimen) for metastatic disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST and ALT no greater than 2 times ULN (no greater than 5 times ULN if liver metastases present) Alkaline phosphatase no greater than 2 times ULN (no greater than 3 times ULN if liver metastases present) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No uncontrolled high blood pressure No unstable angina, symptomatic congestive heart failure, or serious cardiac arrhythmia No New York Heart Association class III or IV heart disease No history of cardiac toxicities with prior fluorouracil and leucovorin calcium No myocardial infarction within the past 6 months Pulmonary: No interstitial pneumonia or extensive and symptomatic fibrosis of the lung Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study No known dihydropyrimidine dehydrogenase deficiency No allergy to platinum-containing drugs No history of intolerance to study anti-emetics (e.g., 5-HT3 antagonists) No known peripheral neuropathy (absence of deep tendon reflexes as sole deficiency allowed) No uncontrolled diabetes No active infection No other active malignancy originating from primary site other than colon or rectum

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics One and only 1 prior chemotherapy regimen for metastatic disease consisting of first-line irinotecan, fluorouracil, and leucovorin calcium (Saltz regimen) Prior adjuvant fluorouracil with leucovorin calcium allowed At least 3 weeks since prior chemotherapy for metastatic disease and recovered No prior adjuvant irinotecan No prior oxaliplatin Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to study lesions unless evidence of progressive disease within the radiotherapy port At least 3 weeks since prior radiotherapy Surgery: See Disease Characteristics At least 4 weeks since prior major surgery and recovered Prior surgical resection of primary tumor or metastases allowed Other: At least 30 days since prior investigational drugs No other concurrent investigational agents No other concurrent anti-cancer therapy No concurrent participation in other investigational trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: Mace L. Rothenberg, MD, FACP, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (134):
- United States (121):
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - Oncology Center at Providence Park, Mobile, Alabama
  - Arizona Clinical Research Center, Tucson, Arizona
  - Arkansas Oncology Associates, P.A., Little Rock, Arkansas
  - Offices of Richard Shapiro, Benjamin Stafford, and Sharon J. Yee, Arcadia, California
  - California Cancer Care, Inc., Greenbrae, California
  - Medical Oncology Internal Medicine, Los Angeles, California
  - Bay Area Tumor Institute, Oakland, California
  - Medical Oncology Care Associates, Orange, California
  - P.M.K. Medical Group, Inc., Oxnard, California
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente - Denver, Denver, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Northwestern Connecticut Oncology-Hematology Associates, Torrington, Connecticut
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Comprehensive Cancer Care Specialists of Boca Raton, Boca Raton, Florida
  - Center for Hematology-Oncology, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - Florida Community Cancer Center, Hudson, Florida
  - North Florida Hematology & Oncology Associates, Jacksonville, Florida
  - Hematology/Oncology Associates, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Office of Thomas A. Marsland, Orange Park, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Office of Barry S. Berman, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Hematology-Oncology Associates, PA, Pensacola, Florida
  - Hematology/Oncology Associates, Port Saint Lucie, Florida
  - Oncology & Hematology Associates of West Broward, Tamarac, Florida
  - Office of Ron D. Schiff, Tampa, Florida
  - Hematology and Oncology Consultants, Titusville, Florida
  - Dreyer Medical Clinic, Aurora, Illinois
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Oncology and Hematology Associates, Greenfield, Indiana
  - Cancer Care Center, New Albany, Indiana
  - Oncology Associates of Cedar Rapids, Cedar Rapids, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Physicians Office, Metairie, Louisiana
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Parker Hughes Cancer Center, Roseville, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - Columbia Comprehensive Cancer Care Clinic, Columbia, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Midwest Oncology Consortium, Kansas City, Missouri
  - Missouri Cancer Care, P.C., Saint Charles, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore Hematology/Oncology Associates, P.C., East Setauket, New York
  - Capitol District Hematology Oncology Associates, P.C., Latham, New York
  - St. Vincents Comprehensive Cancer Center, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Regional Hematology Oncology Associates, Durham, North Carolina
  - Raleigh Hematology/Oncology Associates - Wake Practice, Raleigh, North Carolina
  - Piedmont Hematology-Oncology Associates-Triad, Winston-Salem, North Carolina
  - Hematology Oncology Consultants Inc, Columbus, Ohio
  - Dayton Oncology/Hematology P.A., Dayton, Ohio
  - Naz Medical Center, Midwest City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Oncology/Hematology Associates - Beaver, Beaver, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Erlanger Health Systems, Chattanooga, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - West Clinic, P.C., Memphis, Tennessee
  - Memphis Cancer Center, Memphis, Tennessee
  - St. Thomas Medical Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Lone Star Oncology, Austin, Texas
  - Texas Oncology P.A., Dallas, Texas
  - Center for Oncology Research and Treatment, Medical City Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Texas Cancer Center Southwest, Dallas, Texas
  - Texas Oncology PA (TOPA) at Baylor-Sammons, Dallas, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Texas Oncology, P.A., Garland, Texas
  - South Texas Regional Cancer Centers - McAllen, McAllen, Texas
  - Texas Oncology - Mesquite, Mesqutie, Texas
  - Baptist Health System Cancer Program, San Antonio, Texas
  - San Antonio Tumor and Blood Clinic, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Hematology-Oncology Associates of Frederiksburg, Inc., Fredericksburg, Virginia
  - Virginia Oncology Associates - Newport News, Newport News, Virginia
  - Hematology & Oncology Associates of Virginia, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Advanced Health Care, Milwaukee, Wisconsin
  - UW Cancer Center Wausau Hospital, Wausau, Wisconsin
  - Ivinson Memorial Hospital, Laramie, Wyoming
- Canada (13):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Belleville General Hospital, Belleville, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Notre Dame Hospital, Montreal, Quebec
  - Centre Hospitalier Regional de Rimouski, Rimouski, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan